CLINICAL TRIAL: NCT03469661
Title: Differential Diagnostic of ITP and MDS: a Prospective Study by Next-Generation Flow Cytometry and Cytomorphological Approaches
Brief Title: Differential Diagnostic of Immune ThrombocytoPenia (ITP) and Myelodysplastic Syndrome (MDS)
Status: Completed | Type: Observational
Sponsor: Fundacion CRIS de Investigación para Vencer el Cáncer (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: FCR-PTI-2017-01
Record Dates: First submitted 2018-03-02; First posted 2018-03-19 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Immune Thrombocytopenia; Myelodysplastic Syndromes
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Given a diagnosis of ITP or low-risk MDS, EDTA-anticoagulated bone marrow and peripheral blood aspirates will be obtained per case. A biopsy sample and two unstained blood smears should also be included
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immune Thrombocytopenia Diagnosis
- Myelodysplastic Syndrome Diagnosis

SUMMARY:
Current diagnostic criteria for Immune ThrombocytoPenia (ITP) are mainly based on the presence of low numbers of platelets, excluding other multiple causes of thrombocytopenia, including immunodeficiencies, constitutional or acquired thrombocytopenia, hypersplenism and clonal hematological disorders such as MDS, disorders lymphoproliferative and acute myeloid leukemia (AML), among others. The analysis complementary tests for the diagnosis of ITP include studies basic systematic hematology, together with autoimmune assays and microbiological tests, while the evaluation of bone marrow is limited to elderly patients and/or patients resistant to treatment. Previous research has described the development of Myelodysplastic Syndrome (MDS) in patients with a previous diagnosis of ITP, and even the presence of MDS associated with genetic background. Therefore, it is conceivable fact that a percentage of cases with clinical signs of ITP in the moment of appearance may actually correspond to the first stages of MDS development in which bone marrow cells are not systematically evaluated in the initial presentation.

The anomalous immunophenotypic patterns between multiple compartments of bone marrow cells and peripherally blood (PB) platelets have been characterized through flow cytometry. The flow cytometry currently represents an important complementary tool for diagnosis of MDS that has shown great effectiveness and applicability in the differential diagnosis of non-clonal cytopenias against early MDS and for the detection of stages prior to MDS. Besides, the flow cytometry has made it possible to detect the presence of coexisting features related to MDS in patients with other malignancies hematologic conditions such as multiple myeloma, AML, and lymphocytic leukemia chronic. Therefore, the immunophenotypic analysis of the cells of the bone marrow of patients with ITP at the time of appearance would help to identify the cases that underlie clonal hematopoiesis MDS type. In the present study it is planned a broad characterization immunophenotyping of multiple compartments of bone marrow cells and PB platelets from patients with recently diagnosed ITP and investigate their morphological antecedents, in order to identify those patients who show compatible clonal hematopoietic patterns with MDS evident (or at risk of development), as candidates to receive most appropriate therapeutic methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years old at diagnosis
* Informed consent in writing
* Newly diagnosed primary ITP patients, or
* Newly diagnosed MDS patients

Exclusion Criteria:

* Patients who participated in a interventional thrombopoietin receptor agonists (TPO-RA) clinical trial since TPO-RA treatment initiation
* Patients with secondary immune thrombopenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is estimated that approximately 60 patients will be included in the study, 30 newly diagnosed ITP patients and 30 newly diagnosed MDS cases.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-04-19 (Actual)

PRIMARY OUTCOMES:
Morphological profile | Baseline
  Bone marrow cell compartment profiles
Morphological profile | Baseline
  Peripheral blood platelets profiles
Immunological profile | Baseline
  Bone marrow cell compartment profiles
Immunological profile | Baseline
  Peripheral blood platelets profiles

SECONDARY OUTCOMES:
Immunophenotypic abnormalities | Baseline
  Evaluation of abnormal immunophenotypic profiles
Morphological abnormalities | Baseline
  Evaluation of abnormal morphological profiles.

CONTACTS AND LOCATIONS:
Overall Officials: Tomás González, Principal Investigator — Hospital de Burgos
Locations (6):
- Spain (6):
  - Complejo Hospitalario de A Coruña, A Coruña
  - Hospital de Burgos, Burgos
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria
  - Hospital Ramon y Cajal, Madrid
  - Hospital Regional de Málaga, Málaga
  - Hospital Virgen de la Victoria, Málaga